CLINICAL TRIAL: NCT00755716
Title: Topiramate Alone and in Combination With the Nicotine Patch for Smoking Cessation: A Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Cheryl Oncken, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-114-1; 5M01RR006192 (NIH); K24AA013736 (NIH)
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Dependence
Keywords: nicotine patch; smoking; topiramate
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Sugars; Topiramate; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (sugar pill) (Placebo Comparator): Person receives an inactive placebo
  Interventions: Drug: Placebo (sugar pill)
- Topiramate (Active Comparator): Subjects receive 10 weeks of topiramate with a dosage starting at 25 mg per day. At week two (quit date) subjects increase to 50 mg/day and gradually increase to 200 mg/day for a total time of 10 weeks.
  Interventions: Drug: Topiramate
- Topiramate and Nicotine patch (Active Comparator): Subjects receive 10 weeks of topiramate with a dosage starting at 25 mg per day. At week two (quit date) subjects increase to 50 mg/day and gradually increase to 200 mg/day and one week taper for a total time of 10 weeks. On the quit date (after 2 weeks of Topiramate medication use), subjects also use 21 mg patch for 7 weeks and on week 8 subjects received 14 mg/day for 3 days then 7 mg for 4 days.
  Interventions: Drug: Topiramate; Drug: Nicotine patch

INTERVENTIONS:
Drug: Placebo (sugar pill) — patients receive
  Other Names: sugar pill
  Arms: Placebo (sugar pill)
Drug: Topiramate — 25 mg per day for one week, 50 mg per day for one week, 100 mg per day for one week, 200 mg per day for 5 weeks, then one week taper
  Other Names: topimax
  Arms: Topiramate; Topiramate and Nicotine patch
Drug: Nicotine patch — On the quit date (after 2 weeks of Topiramate medication use), subjects also use 21 mg patch for 7 weeks and on week 8 subjects received 14 mg/day for 3 days then 7 mg for 4 days.
  Other Names: nicoderm
  Arms: Topiramate and Nicotine patch

SUMMARY:
Specific aims:

1. To obtain pilot data on 4-week continuous quit rates associated with 10 weeks of treatment with topiramate or placebo or topiramate plus nicotine patch for smoking cessation.
2. To obtain pilot data on the effects of 10 weeks of topiramate versus placebo versus combination of topiramate plus nicotine patch on nicotine withdrawal symptoms, smoking satisfaction, and adverse effects during smoking cessation.
3. To obtain pilot data on weight gain over 10 weeks with topiramate versus placebo versus combination of topiramate plus nicotine patch for smoking cessation.

DETAILED DESCRIPTION:
This is a 10-week, randomized, double-blind, single-site study of treatment with either: topiramate, or placebo, or topiramate plus nicotine patch. Approximately, 90 subjects ages 18-65 who smoke at least 10 cigarettes per day will be screened for study participation, with the intention of 60 subjects being eligible for randomized treatment (20 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cigarette smoker between the ages of 18 and 65 years inclusive and relatively healthy.
* Subjects must smoke an average of at least 10 cigarettes per day during the past year and during the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.
* BMI > 18kg/in2.
* Subjects must be free of serious or unstable disease within the past 6 months
* Female subjects must be a) postmenopausal for at least two years, or practicing an effective method of birth control (e.g., surgically sterile, prescription oral contraceptives, contraceptive injections, intrauterine device, spermicide with barrier, contraceptive patch, contraceptive ring, male partner sterilization, abstinence and agree to continue abstinence or to use an acceptable method of contraception, as listed above, should sexual activity commence) before entry and throughout the study; have a negative urine pregnancy test at the screening visit. b) agree to avoid pregnancy through 30 days after the last dose of study medication, c) have a negative urine pregnancy test (β-hCG) at screening or baseline and agree to use at least one of the birth control methods as noted in the protocol.
* Subjects must be able to be seen as an outpatient, to be assessed in a clinic setting, and able and willing to comply with all study visits.
* Subjects must be able to provide written consent.
* Subjects must be the only member of the household participating in this study.

Exclusion criteria:

* Subjects who are currently suffering from depression or have been diagnosed with depression or treated with an antidepressant within the past 12 months.
* Subjects who have a past or present history of psychosis, panic disorder, or bipolar disorder.
* Subjects who have severe chronic obstructive pulmonary disease (COPD).4. Subjects who have clinically significant cardiovascular disease in the past 6 months
* Subjects who have clinically significant cardiovascular disease in the past 6 months which includes: myocardial infarction, coronary artery bypass graft CABG), percutaneous transluminal coronary angioplasty (PTCA), severe or unstable angina, serious arrhythmia, and clinically significant ECG conduction abnormalities.
* Subjects who have uncontrolled hypertension or a systolic blood pressure greater than 150 mm Hg or a diastolic blood pressure greater than 95 mm Hg at screening or baseline.
* Subjects who have a history of clinically significant neurological disorders including subjects with seizure disorders, cerebrovascular diseases stroke or transient ischemic attack) and/or progressive or degenerative neurological disorders (e.g., multiple sclerosis) in the past 6 months.
* Subjects who have a history of clinically significant endocrine disorders or gastrointestinal diseases, including insulin dependent diabetes, uncontrolled hyperthyroidism, and active peptic ulcer.
* Subjects who have clinically significant hepatic or renal impairment (e.g., an estimated creatinine clearance <60 mL/min).
* Subjects who have an SGOT (AST) or SGPT (ALT) concentration greater than 1.5 times the upper limit of normal.
* Subjects who have a history of cancer.
* Subjects who are believed to be medically unstable and/or not appropriate for study participation in the opinion of the principal investigator.
* Subjects who have previously been treated with topiramate for any reason and discontinued treatment due to an adverse event or due to a hypersensitivity reaction to topiramate.
* Subjects with evidence or a history of clinically significant allergic reaction.
* Subjects who have an allergy to adhesive tape or a skin disorder that may be exacerbated by nicotine patch.
* Subjects with a history of drug (except nicotine) or alcohol abuse or dependence within the past 12 months.
* Subjects with a positive urine drug screen.
* Subjects that have been enrolled in a study that included topiramate.
* Subjects who have taken or will plan to take another investigational drug within 30 days or 5 half-lives (whichever is longer) before the Baseline visit or within 30 days of study completion.
* Subjects who take or plan to take a concomitant medication that is prohibited by this protocol.
* Subjects who require other medications during the study that might interfere with the evaluation of the study drug (for example, nicotine replacement therapy and bupropion).
* Subjects who used a nicotine replacement product, bupropion, clonidine, or nortriptyline within the past 6 months, or participated in a study with an experimental drug for smoking cessation within the past one year.
* Subjects who intend to use non-cigarette tobacco products (including, for example, pipe tobacco, cigars, snuff, chewing tobacco, etc.) or marijuana during study participation.
* Subjects who intend to donate blood or blood components while receiving study drug or within 1 month of the completion of the study treatment.
* Subjects who are unable and/or unlikely to comprehend and follow the study protocol, which includes a) a subject who, in the investigator's opinion, will be unlikely to commit to the duration of the study, b) a subject who, in the investigator's opinion should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the topiramate package insert.
* Subjects who have lactose intolerance.
* Subjects with a history of glaucoma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Oncken, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Halth Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oncken C, Arias AJ, Feinn R, Litt M, Covault J, Sofuoglu M, Kranzler HR. Topiramate for smoking cessation: a randomized, placebo-controlled pilot study. Nicotine Tob Res. 2014 Mar;16(3):288-96. doi: 10.1093/ntr/ntt141. Epub 2013 Sep 21. PMID 24057996
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- See also: Topiramate for smoking cessation: a randomized, placebo-controlled pilot study — https://www.ncbi.nlm.nih.gov/pubmed/24057996

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Sugar Pill): Person receives an inactive placebo
  Placebo (sugar pill):
- Topiramate: Subjects receive 10 weeks of topiramate with a dosage starting at 25 mg per day. At week two (quit date) subjects increase to 50 mg/day and gradually increase to 200 mg/day and one week taper for a total time of 10 weeks.
Period: Overall Study
Arm/Group | Placebo (Sugar Pill) | Topiramate | Topiramate and Nicotine Patch
Started | 19 | 19 | 19
Completed | 11 | 11 | 16
Not Completed | 8 | 8 | 3
Not completed — Adverse Event | 1 | 4 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 5 | 3 | 1
Not completed — work schedule issues | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Topiramate and Nicotine Patch: Subjects receive 10 weeks of topiramate with a dosage starting at 25 mg per day. At week two (quit date) subjects increase to 50 mg/day and gradually increase to 200 mg/day and one week taper for a total time of 10 weeks.On the quit date (after 2 weeks of Topiramate medication use), subjects also use 21 mg patch for 7 weeks and on week 8 subjects received 14 mg/day for 3 days then 7 mg for 4 days.
- Total: Total of all reporting groups
Arm/Group | Placebo (Sugar Pill) | Topiramate | Topiramate and Nicotine Patch | Total
Number analyzed (Participants) | 19 | 19 | 19 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 19 | 57
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (7.6) | 46.1 (11.1) | 50.1 (9.6) | 47.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 13 | 34
  Male | 8 | 9 | 6 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 19 | 57

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome is 4-week Continuous Quit Rate at the End of Treatment.
Description: The primary efficacy endpoint was CO-confirmed cigarette abstinence during the last 4 weeks of treatment.
Time Frame: weeks 7-10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Sugar Pill) | Topiramate | Topiramate and Nicotine Patch
Number analyzed (Participants) | 19 | 19 | 19
Participants | 1 | 5 | 7

2. Secondary Outcome: MNWS
Description: Minnesota Nicotine Withdrawing Scale
  Scale contains 9 items which are scored 0-4. The total range for the scale is 0-36, where higher scores indicate greater nicotine withdrawal symptoms.
Time Frame: Measured weekly during weeks 7-10 & the mean of weekly measurements is recorded.
Population: Subjects only needed to have an MNWS at one of these time points (weeks 7-10) to be included in the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Sugar Pill) | Topiramate | Topiramate and Nicotine Patch
Number analyzed (Participants) | 16 | 17 | 12
units on a scale | 5.7 (1.3) | 4.9 (1.2) | 6.8 (1.1)

ADVERSE EVENTS:
Time Frame: We assessed adverse events at each weekly visit from randomization through study completion, an average of 10 weeks.
Groups:
- Topiramate & Nicotine Patch: Subjects receive 10 weeks of topiramate with a dosage starting at 25 mg per day. At week two (quit date) subjects increase to 50 mg/day and gradually increase to 200 mg/day and one week taper for a total time of 10 weeks. On the quit date (after 2 weeks of Topiramate medication use), subjects also use 21 mg patch for 7 weeks and on week 8 subjects received 14 mg/day for 3 days then 7 mg for 4 days.
Arm/Group | Placebo (Sugar Pill) | Topiramate | Topiramate & Nicotine Patch
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 16/19 | 17/19 | 18/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Sugar Pill) (N=19) | Topiramate (N=19) | Topiramate & Nicotine Patch (N=19)
Paresthesia (Nervous system disorders) | 0 | 3 | 2
Fatigue (Psychiatric disorders) | 1 | 2 | 5
Loss Of Appetite (Gastrointestinal disorders) | 0 | 1 | 1
Difficulty with Memory (Psychiatric disorders) | 0 | 1 | 2
Weight Loss (Gastrointestinal disorders) | 0 | 1 | 0
Difficulty Concentrating (Psychiatric disorders) | 1 | 2 | 3
Nervousness/agitation/irritablility (Psychiatric disorders) | 4 | 5 | 1
Change in Sense of Taste (General disorders) | 2 | 1 | 2
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 6
Depressed Mood (Psychiatric disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 3
Insomnia (Nervous system disorders) | 0 | 3 | 1
Headache (Nervous system disorders) | 3 | 1 | 3
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Thirst/Dry Mouth (General disorders) | 2 | 1 | 3
Nausea/Vomiting (Gastrointestinal disorders) | 2 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Fever (General disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes